CLINICAL TRIAL: NCT01430559
Title: A DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER, PARALLEL GROUP STUDY OF THE EFFECT OF MELOXICAM IN MAINLAND CHINESE SUBJECTS WITH OSTEOARTHRITIS (OA) OF THE KNEE
Brief Title: Effect Of Meloxicam Versus Placebo In Mainland Chinese Patients With Osteoarthritis Of The Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A9001449
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Validation of the WOMAC in Chinese subjects with osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Meloxicam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meloxicam (Other)
  Interventions: Drug: Meloxicam
- Placebo (Placebo Comparator): 2 Placebo capsules once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meloxicam — 7.5mg x2 once a day for 12 weeks
  Other Names: Mobic
  Arms: Meloxicam
Drug: Placebo — Study subjects will be randomized to two treatment groups: one with Meloxicam 7.5 mgx2 once a day and another one with placebo. The duration of the interventional treatment is 12 weeks.
  Arms: Placebo

SUMMARY:
This study is to validate the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) tool in mainland Chinese patients with osteoarthritis of the knee . This study will also evaluate the effects of Mobic versus placebo on reducing the symptoms of osteoarthritis in this population.

DETAILED DESCRIPTION:
To validate culturally the WOMAC tool in mainland China and observe the different response of meloxicam and placebo in a patient population with osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet the following criteria to be eligible for Randomization into this study:

* Male or female Chinese subjects, 18-75 years of age;
* Subjects must have a diagnosis of OA of the index knee based on American College of Rheumatology criteria with X ray confirmation (a Kellgren Lawrence x ray grade of greater than or equal to 2) (Kellgren J. & Lawrence J, 1957)
* Subjects must have have an NRS and a WOMAC pain sub scale score of 4 at Screening and at Baseline based on four daily diary entries

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* History of other disease that may involve the index (painful) knee including inflammatory joint diseases or have had recent surgical intervention on the knee.
* Diagnosed as having or has been treated for esophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to receiving the first dose of study medication. History of or active gastrointestinal disease (eg, inflammatory bowel disease), a chronic or acute renal or hepatic disorder, or a significant coagulation defect.
* Signs and symptoms of clinically significant cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2011-10-24 (Actual); Primary Completion 2013-03-27 (Actual); Study Completion 2013-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- China (25):
  - Anhui Province Hospital, Hefei, Anhui
  - The Third Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou Medical Collage, Shantou, Guangdong
  - Rheumatology Department, The first Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Rheumatology Department, The First Hospital of China Medical University, Shenyang, Liaoning
  - QiLu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital/Orthopaedics, Liaocheng, Shandong
  - Department of Immunology and Rheumatology, Qingdao Municipal Hospital, Qingdao, Shandong
  - Department of Immunology and Rheumatology,Qingdao Municipal Hospital, Qingdao, Shandong
  - Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Department of Orthopedics, West China Hospital of Sichuan University, Chengdu, Sichuan
  - Department of Rheumatology and Immunology,West China Hospital of Sichuan University, Chengdu, Sichuan
  - Department of Rheumatology and Immunology, Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Rheumatology, Chengdu, Sichuan
  - China-Japan Friendship Hospital/Rheumatology Department, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Li Zhanguo, Beijing
  - Rheumatology and Immunology Department, Xuanwu Hospital Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Orthopaedics, Beijing
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Rheumatology and Immunology Department, Shanghai Changzheng Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Rheumatology Department, Shanghai
  - Department of Infectious Diseases & Immunology, Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001449&StudyName=Effect%20Of%20Meloxicam%20Versus%20Placebo%20In%20Mainland%20Chinese%20Patients%20With%20Osteoarthritis%20Of%20The%20Knee%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 centers in mainland China recruited study participants, starting from 24 Oct 2011 to 14 Dec 2012.
Pre-assignment Details: This study comprised of a Screening Period prior to Treatment Period. During Screening, 52 healthy participants and 356 participants with osteoarthritis (OA) were included in validation analysis set (total enrollment=408), 293 out of the 356 OA participants were assigned randomized to treatment, and 6 of these randomized participants did not receive actual treatment.
Groups:
- Placebo: Participants were randomized to placebo treatment group at Baseline and received matching placebo (2 capsules once daily) for 12 weeks.
- Meloxicam 15 mg: Participants were randomized to meloxicam treatment group at Baseline and received meloxicam 7.5 milligram (mg) × 2 once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Meloxicam 15 mg
Started | 146 | 147
Treated | 143 | 144
Completed | 126 | 135
Not Completed | 20 | 12
Not completed — Adverse Event | 7 | 3
Not completed — Entry criteria not met | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Medication error | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 3 | 3
Not completed — Randomized, Not Treated | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Meloxicam 15 mg | Total
Number analyzed (Participants) | 143 | 144 | 287
Age, Customized [Count of Participants; unit: Participants]
  26 to 35 years | 1 | 1 | 2
  36 to 45 years | 4 | 12 | 16
  46 to 55 years | 43 | 44 | 87
  56 to 65 years | 61 | 60 | 121
  66 to 75 years | 34 | 27 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 122 | 228
  Male | 37 | 22 | 59

OUTCOME MEASURES:

1. Primary Outcome: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Total and the 3 Subscales Scores (Pain, Stiffness and Physical Function) at Screening 1 by Using a Paper Worksheet and a Personalized Electronic LogPad System (E-diary)
Description: The WOMAC has 3 subscales: WOMAC pain subscale, WOMAC stiffness subscale and WOMAC physical function subscale, which are comprised of 5, 2 and 17 questions regarding the amount of pain and stiffness experienced in the index knee, and degree of difficulty in doing daily tasks, respectively in the past 48 hours. The WOMAC subscale scores range from 0 to 10 with higher scores indicating higher pain, more stiffness and worse function respectively for pain, stiffness and physical function subscales. The WOMAC subscale scores were calculated as the mean of the scores from the individual questions. The WOMAC total score was the sum of scores from the 5, 2 and 17 questions respectively on pain, stiffness and physical function subscales. WOMAC total score ranged from 0 to 240, where higher scores indicated worse health condition.
Time Frame: Screening 1 (Visit 1: Days -21 to -14)
Population: Validation Analysis Set (VAS) - all OA participants who were non-screen failure at Visit 1 (Screening 1) and returned for Visit 2 (Screening 2); and all enrolled healthy participants. Here, n=number of evaluable participants for each specific category.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OA Participants: Participants with OA who responded to the WOMAC questionnaire.
- Healthy Participants: Healthy participants who responded to the WOMAC questionnaire.
Arm/Group | OA Participants | Healthy Participants
Number analyzed (Participants) | 356 | 52
units on a scale
  Pain subscale (paper worksheet): number analyzed (Participants) | 356 | 0
  Pain subscale (paper worksheet) | 5.7 (1.47) |
  Stiffness subscale (paper worksheet): number analyzed (Participants) | 356 | 0
  Stiffness subscale (paper worksheet) | 5.3 (1.94) |
  Physical function subscale (paper worksheet): number analyzed (Participants) | 356 | 0
  Physical function subscale (paper worksheet) | 5.7 (1.56) |
  Total (paper worksheet): number analyzed (Participants) | 356 | 0
  Total (paper worksheet) | 135.9 (35.59) |
  Pain subscale (e-dary) | 5.7 (1.47) | 0.1 (0.22)
  Stiffness subscale (e-diary) | 5.3 (2.00) | 0.1 (0.31)
  Physical function subscale (e-diary) | 5.7 (1.56) | 0.0 (0.14)
  Total (e-diary) | 136.0 (35.92) | 0.8 (3.66)

2. Primary Outcome: WOMAC Total and the 3 Subscales Scores (Pain, Stiffness and Physical Function) at Screening 2 by Using E-diary
Description: as for outcome 1
Time Frame: Screening 2 (Visit 2: Days -14 to -10)
Population: VAS: all OA participants who were non-screen failure at Visit 1 (Screening 1) and returned for Visit 2 (Screening 2).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OA Participants
Number analyzed (Participants) | 356
units on a scale
  Pain subscale score | 5.6 (1.46)
  Stiffness subscale score | 5.4 (1.76)
  Physical function subscale score | 5.8 (1.52)
  Total score | 136.6 (35.38)

3. Primary Outcome: WOMAC Total and the 3 Subscales Scores (Pain, Stiffness and Physical Function) at Baseline by Using E-diary
Description: as for outcome 1
Time Frame: Baseline (Day 1)
Population: FAS: all randomized participants who received at least 1 dose of study medication, number of participants analyzed=number of participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 139 | 139
units on a scale
  Pain subscale score | 6.0 (1.29) | 6.0 (1.32)
  Stiffness subscale score | 5.7 (1.56) | 5.6 (1.65)
  Physical function subscale score | 6.1 (1.32) | 6.1 (1.22)
  Total score | 145.0 (31.05) | 144.8 (29.57)

4. Primary Outcome: WOMAC Total and the 3 Subscales Scores (Pain, Stiffness and Physical Function) at Week 12 by Using E-diary
Description: as for outcome 1
Time Frame: Visit 8 (Week 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 101 | 119
units on a scale
  Pain subscale score | 4.4 (2.05) | 3.6 (1.90)
  Stiffness subscale score | 4.2 (2.26) | 3.5 (1.96)
  Physical function subscale score | 4.5 (2.08) | 3.7 (1.87)
  Total score | 106.6 (49.70) | 88.7 (44.45)

5. Primary Outcome: Change From Baseline in WOMAC Pain Subscale Scores at Week 12
Description: WOMAC pain subscale is comprised of 5 questions regarding the amount of pain experienced in the index knee in the past 48 hours. The WOMAC pain subscale scores range from 0 to 10 with higher scores indicating higher pain. The WOMAC pain subscale score was calculated as the mean of the scores from the individual questions.
Time Frame: Baseline and Week 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using Baseline Observation Carried Forward (BOCF) imputation method, number of participants analyzed=number of participants evaluable for the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 139 | 139
units on a scale | -1.24 [-1.71 to -0.77] | -2.06 [-2.53 to -1.58]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value and 95% confidence interval for least squares mean difference were calculated from analysis of covariance (ANCOVA, repeated measures) model with baseline value and treatment group as fixed effects, and study site as a random effect; Least Squares Mean Difference = -0.82, 95% CI 2-sided [-1.20 to -0.43], Standard Error of Mean 0.19

6. Secondary Outcome: Change From Baseline in WOMAC Subscale and Average Scores at Weeks 2, 4, 8 and 12
Description: The WOMAC has 3 subscales: WOMAC pain subscale, WOMAC stiffness subscale and WOMAC physical function subscale, which are comprised of 5, 2 and 17 questions regarding the amount of pain and stiffness experienced in the index knee, and degree of difficulty in doing daily tasks, respectively in the past 48 hours. The WOMAC subscale scores range from 0 to 10 with higher scores indicating higher pain, more stiffness and worse function respectively for pain, stiffness and physical function subscales. The WOMAC subscale scores were calculated as the mean of the scores from the individual questions. Change from baseline was calculated for each WOMAC subscale (pain, stiffness, physical function) and WOMAC average score.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using BOCF imputation method, number of participants analyzed=number of participants evaluable for the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 139 | 139
units on a scale
  Pain subscale (Week 2) | -0.76 [-1.15 to -0.36] | -1.12 [-1.52 to -0.73]
  Pain subscale (Week 4) | -1.18 [-1.60 to -0.76] | -1.53 [-1.95 to -1.11]
  Pain subscale (Week 8) | -1.31 [-1.74 to -0.87] | -1.82 [-2.26 to -1.39]
  Pain subscale (Week 12) | -1.24 [-1.71 to -0.77] | -2.06 [-2.53 to -1.58]
  Stiffness subscale (Week 2) | -0.78 [-1.16 to -0.39] | -1.11 [-1.49 to -0.72]
  Stiffness subscale (Week 4) | -1.14 [-1.58 to -0.71] | -1.34 [-1.78 to -0.90]
  Stiffness subscale (Week 8) | -1.23 [-1.66 to -0.79] | -1.70 [-2.14 to -1.25]
  Stiffness subscale (Week 12) | -1.20 [-1.67 to -0.72] | -1.86 [-2.34 to -1.39]
  Physical function subscale (Week 2) | -0.77 [-1.19 to -0.36] | -1.21 [-1.63 to -0.80]
  Physical function subscale (Week 4) | -1.18 [-1.62 to -0.75] | -1.53 [-1.96 to -1.09]
  Physical function subscale (Week 8) | -1.31 [-1.74 to -0.88] | -1.82 [-2.26 to -1.38]
  Physical function subscale (Week 12) | -1.25 [-1.73 to -0.77] | -2.06 [-2.54 to -1.58]
  Average score (Week 2) | -0.77 [-1.15 to -0.39] | -1.15 [-1.54 to -0.77]
  Average score (Week 4) | -1.17 [-1.60 to -0.75] | -1.47 [-1.90 to -1.04]
  Average score (Week 8) | -1.29 [-1.71 to -0.86] | -1.78 [-2.22 to -1.35]
  Average score (Week 12) | -1.23 [-1.70 to -0.76] | -2.00 [-2.47 to -1.52]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Pain subscale (Week 2); Test type: Superiority or Other; p = 0.0103, ANCOVA — P-value and 95% confidence interval for least squares mean difference were calculated from ANCOVA (repeated measures) model with baseline value and treatment group as fixed effects, and study site as a random effect; Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.65 to -0.09], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Pain subscale (Week 4); Test type: Superiority or Other; p = 0.0295, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.35, 95% CI 2-sided [-0.67 to -0.04], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Pain subscale (Week 8); Test type: Superiority or Other; p = 0.0041, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.52, 95% CI 2-sided [-0.87 to -0.17], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Pain subscale (Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.82, 95% CI 2-sided [-1.20 to -0.43], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Placebo vs Meloxicam 15 mg; Stiffness subscale (Week 2); Test type: Superiority or Other; p = 0.0369, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.64 to -0.02], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Placebo vs Meloxicam 15 mg; Stiffness subscale (Week 4); Test type: Superiority or Other; p = 0.2642, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.20, 95% CI 2-sided [-0.54 to 0.15], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs Meloxicam 15 mg; Stiffness subscale (Week 8); Test type: Superiority or Other; p = 0.0140, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-0.84 to -0.10], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Placebo vs Meloxicam 15 mg; Stiffness subscale (Week 12); Test type: Superiority or Other; p = 0.0009, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.67, 95% CI 2-sided [-1.06 to -0.28], Standard Error of Mean 0.20
Statistical Analysis 9: Comparison: Placebo vs Meloxicam 15 mg; Physical function subscale (Week 2); Test type: Superiority or Other; p = 0.0017, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.44, 95% CI 2-sided [-0.72 to -0.17], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Placebo vs Meloxicam 15 mg; Physical function subscale (Week 4); Test type: Superiority or Other; p = 0.0328, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.35, 95% CI 2-sided [-0.66 to -0.03], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Meloxicam 15 mg; Physical function subscale (Week 8); Test type: Superiority or Other; p = 0.0043, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.51, 95% CI 2-sided [-0.86 to -0.16], Standard Error of Mean 0.18
Statistical Analysis 12: Comparison: Placebo vs Meloxicam 15 mg; Physical function subscale (Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.81, 95% CI 2-sided [-1.19 to -0.43], Standard Error of Mean 0.19
Statistical Analysis 13: Comparison: Placebo vs Meloxicam 15 mg; Average score (Week 2); Test type: Superiority or Other; p = 0.0051, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.38, 95% CI 2-sided [-0.65 to -0.12], Standard Error of Mean 0.13
Statistical Analysis 14: Comparison: Placebo vs Meloxicam 15 mg; Average score (Week 4); Test type: Superiority or Other; p = 0.0593, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.61 to 0.01], Standard Error of Mean 0.16
Statistical Analysis 15: Comparison: Placebo vs Meloxicam 15 mg; Average score (Week 8); Test type: Superiority or Other; p = 0.0046, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.50, 95% CI 2-sided [-0.84 to -0.16], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Meloxicam 15 mg; Average score (Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.76, 95% CI 2-sided [-1.14 to -0.39], Standard Error of Mean 0.19

7. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Items at Weeks 2, 4, 8 and 12
Description: WOMAC pain subscale is comprised of 5 questions regarding the amount of pain experienced in the index knee in the past 48 hours. The WOMAC pain subscale scores range from 0 to 10 with higher scores indicating higher pain. Change from baseline in two of the WOMAC pain subscale items: pain when walking on a flat surface, and pain when going up or down stairs were calculated.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 139 | 139
units on a scale
  Walking on flat surface (Week 2) | -0.51 [-0.92 to -0.10] | -1.13 [-1.54 to -0.71]
  Walking on flat surface (Week 4) | -1.04 [-1.50 to -0.59] | -1.61 [-2.07 to -1.15]
  Walking on flat surface (Week 8) | -1.17 [-1.63 to -0.71] | -1.87 [-2.33 to -1.41]
  Walking on flat surface (Week 12) | -1.05 [-1.53 to -0.56] | -1.97 [-2.46 to -1.48]
  Going up or down stairs (Week 2) | -1.00 [-1.40 to -0.60] | -1.35 [-1.75 to -0.94]
  Going up or down stairs (Week 4) | -1.34 [-1.76 to -0.93] | -1.74 [-2.16 to -1.32]
  Going up or down stairs (Week 8) | -1.53 [-2.00 to -1.07] | -2.09 [-2.55 to -1.62]
  Going up or down stairs (Week 12) | -1.34 [-1.83 to -0.86] | -2.43 [-2.91 to -1.94]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Walking on flat surface (Week 2); Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.62, 95% CI 2-sided [-0.94 to -0.30], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Walking on flat surface (Week 4); Test type: Superiority or Other; p = 0.0015, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.57, 95% CI 2-sided [-0.92 to -0.22], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Walking on flat surface (Week 8); Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-1.08 to -0.32], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Walking on flat surface (Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.93, 95% CI 2-sided [-1.34 to -0.51], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Placebo vs Meloxicam 15 mg; Going up or down stairs (Week 2); Test type: Superiority or Other; p = 0.0363, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.35, 95% CI 2-sided [-0.67 to -0.02], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Placebo vs Meloxicam 15 mg; Going up or down stairs (Week 4); Test type: Superiority or Other; p = 0.0311, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.75 to -0.04], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs Meloxicam 15 mg; Going up or down stairs (Week 8); Test type: Superiority or Other; p = 0.0057, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.55, 95% CI 2-sided [-0.94 to -0.16], Standard Error of Mean 0.20
Statistical Analysis 8: Comparison: Placebo vs Meloxicam 15 mg; Going up or down stairs (Week 12); Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -1.08, 95% CI 2-sided [-1.52 to -0.64], Standard Error of Mean 0.22

8. Secondary Outcome: Percentage of Participants With Cumulative Reduction From Baseline in WOMAC Pain Subscale at Week 12
Description: WOMAC pain subscale is comprised of 5 questions regarding the amount of pain experienced in the index knee in the past 48 hours. The WOMAC pain subscale scores range from 0 to 10 with higher scores indicating higher pain. The WOMAC pain subscale score was calculated as the mean of the scores from the individual questions. WOMAC pain subscale response rates at Week 12 were shown for the reductions from Baseline of greater than (>) 0%, 10% to 90% (in steps of 10%).
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 139 | 139
percentage of participants
  >0% reduction | 53.1 | 75.7
  Greater than or equal to (>=) 10% reduction | 46.2 | 67.4
  >=20% reduction | 37.1 | 58.3
  >=30% reduction | 29.4 | 49.3
  >=40% reduction | 22.4 | 43.8
  >=50% reduction | 16.1 | 34.0
  >=60% reduction | 10.5 | 24.3
  >=70% reduction | 7.7 | 12.5
  >=80% reduction | 4.2 | 6.3
  >=90% reduction | 2.1 | 3.5

9. Secondary Outcome: Percentage of Participants With at Least 30% and 50% Reduction From Baseline in the WOMAC Pain Subscale at Weeks 2, 4, 8, and 12
Description: as for outcome 5
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using BOCF imputation method, number of participants analyzed=number of participants evaluable for the outcome measure, including the 9 participants (4 placebo, 5 meloxicam) who had missing baseline WOMAC data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 143 | 144
percentage of participants
  >=30% reduction (Week 2) | 17.48 | 22.92
  >=30% reduction (Week 4) | 30.07 | 36.81
  >=30% reduction (Week 8) | 34.97 | 45.14
  >=30% reduction (Week 12) | 29.37 | 49.31
  >=50% reduction (Week 2) | 4.90 | 9.03
  >=50% reduction (Week 4) | 9.09 | 14.58
  >=50% reduction (Week 8) | 13.29 | 24.31
  >=50% reduction (Week 12) | 16.08 | 34.03
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; >=30% reduction (Week 2); Test type: Superiority or Other; p = 0.2373, Regression, Logistic — P-value and 95% confidence interval for odds ratio were calculated from logistic regression model (including baseline value and treatment group as factors) for binary data for comparison of meloxicam group versus placebo; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.79 to 2.55]
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; >=30% reduction (Week 4); Test type: Superiority or Other; p = 0.2069, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.84 to 2.26]
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; >=30% reduction (Week 8); Test type: Superiority or Other; p = 0.0680, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.97 to 2.53]
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; >=30% reduction (Week 12); Test type: Superiority or Other; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.47 to 3.94]
Statistical Analysis 5: Comparison: Placebo vs Meloxicam 15 mg; >=50% reduction (Week 2); Test type: Superiority or Other; p = 0.1736, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.75 to 5.01]
Statistical Analysis 6: Comparison: Placebo vs Meloxicam 15 mg; >=50% reduction (Week 4); Test type: Superiority or Other; p = 0.1496, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.82 to 3.59]
Statistical Analysis 7: Comparison: Placebo vs Meloxicam 15 mg; >=50% reduction (Week 8); Test type: Superiority or Other; p = 0.0171, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.14 to 3.93]
Statistical Analysis 8: Comparison: Placebo vs Meloxicam 15 mg; >=50% reduction (Week 12); Test type: Superiority or Other; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.57 to 4.89]

10. Secondary Outcome: Change From Baseline in Patient Global Assessment of Osteoarthritis (PGAO) at Weeks 2, 4, 8 and 12
Description: PGAO questionnaire ("Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?") was comprised of 5 scores with 1=very good to 5=very poor, where higher grades indicated more effect of osteoarthritis.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 140 | 139
units on a scale
  Week 2 | -0.27 [-0.39 to -0.15] | -0.45 [-0.57 to -0.33]
  Week 4 | -0.37 [-0.50 to -0.23] | -0.53 [-0.66 to -0.39]
  Week 8 | -0.34 [-0.46 to -0.23] | -0.52 [-0.64 to -0.40]
  Week 12 | -0.43 [-0.58 to -0.28] | -0.62 [-0.78 to -0.47]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Week 2; Test type: Superiority or Other; p = 0.0027, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.31 to -0.07], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Week 4; Test type: Superiority or Other; p = 0.0308, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-0.30 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Week 8; Test type: Superiority or Other — P-value and 95% confidence interval for least squares mean difference were calculated from ANCOVA (repeated measures) model with baseline value and treatment group as fixed effects, and study site as a random effect; p = 0.0060, ANCOVA; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-0.31 to -0.05], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Week 12; Test type: Superiority or Other; p = 0.0076, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.20, 95% CI 2-sided [-0.34 to -0.05], Standard Error of Mean 0.07

11. Secondary Outcome: Percentage of Participants With >=2 Points Improvement in PGAO From Baseline at Weeks 2, 4, 8, and 12
Description: PGAO questionnaire ("Considering all the ways your osteoarthritis in your knee affects you, how are you doing today?") was comprised of 5 grades with 1=very good to 5=very poor, where higher grades indicated more effect of osteoarthritis. The treatment response of an improvement of >=2 points from Baseline in PGAO were summarized.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using BOCF imputation method, number of participants analyzed=number of participants evaluable for the outcome measure, including the 8 participants (3 placebo, 5 meloxicam) who had missing baseline PGAO data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 143 | 144
percentage of participants
  Week 2 | 2.80 | 4.86
  Week 4 | 6.29 | 11.81
  Week 8 | 5.59 | 6.25
  Week 12 | 8.39 | 13.19
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Week 2; Test type: Superiority or Other; p = 0.2843, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.53 to 8.50]
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Week 4; Test type: Superiority or Other; p = 0.1050, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.86 to 4.87]
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Week 8; Test type: Superiority or Other; p = 0.7861, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.40 to 3.32]
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Week 12; Test type: Superiority or Other; p = 0.1873, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.77 to 3.78]

12. Secondary Outcome: Change From Baseline in Short-Form 36 Health Survey (SF-36) Domain Scores and Component Scores at Week 12
Description: The SF-36 is a self-administered questionnaire that measures each of the following 8 health domains: physical functioning, role limitations due to physical problems (role-physical), social functioning, bodily pain, mental health, role limitations due to emotional problems (role-emotional), vitality, and general health perception. There are also 2 component scores derived from the 8 subscale scores: physical component summary (including physical functioning, role-physical, bodily pain and general health) and mental component summary (including vitality, social functioning, role-emotional and mental health). Each SF-36 domain and component summary score ranges from 0 to 100, higher scores reflect better participant health status.
Time Frame: Baseline and Week 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using BOCF imputation method, number of participants analyzed=number of participants evaluable for the outcome measure, n=number of evaluable participants for each specific SF-36 domain.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 143 | 144
units on a scale
  General health: number analyzed (Participants) | 141 | 143
  General health | 4.60 [1.93 to 7.28] | 5.98 [3.29 to 8.67]
  Physical functioning: number analyzed (Participants) | 141 | 142
  Physical functioning | 6.95 [3.73 to 10.16] | 12.88 [9.65 to 16.12]
  Role physical: number analyzed (Participants) | 141 | 143
  Role physical | 5.79 [1.74 to 9.84] | 13.95 [9.89 to 18.02]
  Bodily pain: number analyzed (Participants) | 141 | 143
  Bodily pain | 7.51 [4.44 to 10.58] | 14.87 [11.78 to 17.96]
  Vitality: number analyzed (Participants) | 141 | 143
  Vitality | 5.03 [2.56 to 7.50] | 7.08 [4.61 to 9.55]
  Social functioning: number analyzed (Participants) | 141 | 143
  Social functioning | 6.06 [2.60 to 9.51] | 12.02 [8.55 to 15.49]
  Role emotional: number analyzed (Participants) | 141 | 143
  Role emotional | 4.65 [0.26 to 9.04] | 10.52 [6.11 to 14.93]
  Mental health: number analyzed (Participants) | 141 | 143
  Mental health | 4.50 [2.13 to 6.87] | 5.07 [2.71 to 7.43]
  Mental component aggregate: number analyzed (Participants) | 141 | 142
  Mental component aggregate | 2.19 [0.74 to 3.65] | 3.14 [1.67 to 4.60]
  Physical component aggregate: number analyzed (Participants) | 141 | 142
  Physical component aggregate | 2.65 [1.36 to 3.94] | 5.21 [3.92 to 6.51]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; General health; Test type: Superiority or Other; p = 0.3738, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 1.38, 95% CI 2-sided [-1.67 to 4.42], Standard Error of Mean 1.55
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Physical functioning; Test type: Superiority or Other; p = 0.0028, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 5.94, 95% CI 2-sided [2.07 to 9.80], Standard Error of Mean 1.96
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Role physical; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 8.16, 95% CI 2-sided [3.95 to 12.38], Standard Error of Mean 2.14
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Bodily pain; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 7.36, 95% CI 2-sided [4.10 to 10.63], Standard Error of Mean 1.66
Statistical Analysis 5: Comparison: Placebo vs Meloxicam 15 mg; Vitality; Test type: Superiority or Other; p = 0.2124, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 2.05, 95% CI 2-sided [-1.18 to 5.27], Standard Error of Mean 1.64
Statistical Analysis 6: Comparison: Placebo vs Meloxicam 15 mg; Social functioning; Test type: Superiority or Other; p = 0.0050, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 5.96, 95% CI 2-sided [1.82 to 10.10], Standard Error of Mean 2.10
Statistical Analysis 7: Comparison: Placebo vs Meloxicam 15 mg; Role emotional; Test type: Superiority or Other; p = 0.0093, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 5.87, 95% CI 2-sided [1.46 to 10.28], Standard Error of Mean 2.24
Statistical Analysis 8: Comparison: Placebo vs Meloxicam 15 mg; Mental health; Test type: Superiority or Other; p = 0.7274, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 0.57, 95% CI 2-sided [-2.66 to 3.81], Standard Error of Mean 1.64
Statistical Analysis 9: Comparison: Placebo vs Meloxicam 15 mg; Mental component aggregate; Test type: Superiority or Other; p = 0.2819, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 0.94, 95% CI 2-sided [-0.78 to 2.67], Standard Error of Mean 0.88
Statistical Analysis 10: Comparison: Placebo vs Meloxicam 15 mg; Physical component aggregate; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = 2.57, 95% CI 2-sided [1.27 to 3.86], Standard Error of Mean 0.66

13. Secondary Outcome: Percentage of Participants With Change From Baseline in EuroQoL-5 Domains (EQ-5D) Level at Week 12
Description: The EQ-5D is a generic measure of health related quality of life. The EQ-5D has 5 items that assess the level of difficulty (none [score of 1], some/moderate [score of 2], extreme [score of 3]) respondents report for 5 health status domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The change from Baseline (decrease by 2, 1, 0, -1 and -2) at Week 12 in each of the 5 health status domains were summarized.
Time Frame: Baseline and Week 12
Population: FAS: all randomized participants who received at least 1 dose of study medication using BOCF imputation method, number of participants analyzed=number of participants evaluable for the outcome measure, including the 12 participants (5 placebo, 7 meloxicam) who had missing baseline EQ-5D data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 143 | 144
percentage of participants
  Mobility (decrease by 2) | 0 | 0
  Mobility (decrease by 1) | 2.8 | 0.7
  Mobility (decrease by 0) | 79.7 | 66.0
  Mobility (decrease by -1) | 14.0 | 28.5
  Mobility (decrease by -2) | 0 | 0
  Self-care (decrease by 2) | 0 | 0
  Self-care (decrease by 1) | 3.5 | 4.2
  Self-care (decrease by 0) | 67.8 | 55.6
  Self-care (decrease by -1) | 25.2 | 35.4
  Self-care (decrease by -2) | 0 | 0
  Usual activities (decrease by 2) | 0 | 0
  Usual activities (decrease by 1) | 0.7 | 2.8
  Usual activities (decrease by 0) | 81.1 | 63.2
  Usual activities (decrease by -1) | 14.7 | 29.2
  Usual activities (decrease by -2) | 0 | 0
  Pain/discomfort (decrease by 2) | 0 | 0
  Pain/discomfort (decrease by 1) | 2.1 | 2.1
  Pain/discomfort (decrease by 0) | 77.6 | 67.4
  Pain/discomfort (decrease by -1) | 15.4 | 25.0
  Pain/discomfort (decrease by -2) | 1.4 | 0.7
  Anxiety/depression (decrease by 2) | 0.7 | 0
  Anxiety/depression (decrease by 1) | 7.7 | 6.3
  Anxiety/depression (decrease by 0) | 72.0 | 67.4
  Anxiety/depression (decrease by -1) | 14.7 | 20.8
  Anxiety/depression (decrease by -2) | 1.4 | 0.7
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Mobility; Test type: Superiority or Other; p = 0.0014, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.45 to 4.66]
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Self-care; Test type: Superiority or Other; p = 0.1080, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.91 to 2.48]
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Usual activities; Test type: Superiority or Other; p = 0.0119, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.17 to 3.62]
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Pain/discomfort; Test type: Superiority or Other; p = 0.0887, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.93 to 2.83]
Statistical Analysis 5: Comparison: Placebo vs Meloxicam 15 mg; Anxiety/depression; Test type: Superiority or Other; p = 0.2466, Regression, Logistic — [p-value comment as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.80 to 2.33]

14. Secondary Outcome: Change From Baseline in Weekly Average Pain Score in the Index Knee Using 11-point Numeric Rating Scale (NRS) at Weeks 2, 4, 8 and 12
Description: Daily average knee pain was assessed with an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated worse pain. The participants described their pain in the index knee during the past 24 hours by choosing the appropriate number from 0 to 10.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Meloxicam 15 mg
Number analyzed (Participants) | 141 | 143
units on a scale
  Week 2 | -0.67 [-1.00 to -0.34] | -0.97 [-1.30 to -0.64]
  Week 4 | -1.11 [-1.51 to -0.70] | -1.42 [-1.83 to -1.01]
  Week 8 | -1.31 [-1.78 to -0.85] | -1.76 [-2.22 to -1.29]
  Week 12 | -1.43 [-1.94 to -0.91] | -2.06 [-2.57 to -1.55]
Statistical Analysis 1: Comparison: Placebo vs Meloxicam 15 mg; Week 2; Test type: Superiority or Other; p = 0.0367, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.58 to -0.02], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Meloxicam 15 mg; Week 4; Test type: Superiority or Other; p = 0.0652, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.32, 95% CI 2-sided [-0.65 to 0.02], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs Meloxicam 15 mg; Week 8; Test type: Superiority or Other; p = 0.0200, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.44, 95% CI 2-sided [-0.81 to -0.07], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Placebo vs Meloxicam 15 mg; Week 12; Test type: Superiority or Other; p = 0.0016, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.63, 95% CI 2-sided [-1.02 to -0.24], Standard Error of Mean 0.20

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what are presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- OA Participants Not Randomized: OA participants in VAS who were not randomized to placebo or meloxicam treatment.
- OA Participants Randomized But Not Treated: OA participants who were randomized but did not receive actual placebo or meloxicam treatment.
- Healthy Participants: Healthy participants who were included in validation part of the study.
Arm/Group | Placebo | Meloxicam 15 mg | OA Participants Not Randomized | OA Participants Randomized But Not Treated | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 2/143 | 0/144 | 0/63 | 0/6 | 0/52
Other Adverse Events (participants affected / at risk) | 0/143 | 0/144 | 0/63 | 0/6 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Meloxicam 15 mg (N=144) | OA Participants Not Randomized (N=63) | OA Participants Randomized But Not Treated (N=6) | Healthy Participants (N=52)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.